CLINICAL TRIAL: NCT04082429
Title: Efficacy and Safety of Concizumab Prophylaxis in Patients With Haemophilia A or B Without Inhibitors
Brief Title: Research Study to Look at How Well the Drug Concizumab Works in Your Body if You Have Haemophilia Without Inhibitors
Acronym: explorer8
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7415-4307; U1111-1225-9722 (Other: World Health Organization (WHO)); 2018-004891-36 (Registry Identifier: European Medicines Agency (EudraCT))
Expanded Access: NCT04921956 (Available)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Haemophilia A Without Inhibitors; Haemophilia B Without Inhibitors
MeSH Terms: interventions — concizumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to concizumab PPX/no PPX/ assigned into non-randomised arms, based on treatment before trial. Upon restart, patients randomised to arms 1/2 before pause will enter arm 4. Patients allocated to arms 3 & 4 before pause will re-enter initially allocated arm. Randomisation into arms 1/2 will be restarted with new patients. Main part is completed when patient completed 24 wks (excluding screening) in arm 1 or 32 wks (excluding screening) in arms 2-4. After main part, patients will have offer to continue in extension (ext.) part and receive treatment with product until concizumab is commercially available in their countries or until 31-Dec-2027 at latest. Patients will be in the extension part for up to 345 weeks (arms 2-4) or up to 353 weeks (arm 1). Patient will receive last dose at home on day prior to visit 26a. Follow-up part will start on visit 26a and lasts for 7 wks and include reporting of bleeding episodes until visit 27a.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: No prophylaxis (PPX) (Experimental): Haemophilia A (HA) and haemophilia B (HB) patients, previously treated on-demand, will be randomised 1:2 to no prophylaxis versus concizumab prophylaxis. In the extension phase, this group will receive treatment with concizumab.
  Interventions: Drug: Concizumab
- Arm 2: Concizumab prophylaxis (Experimental): HA and HB patients, previously treated on-demand, will be randomised 1:2 to no prophylaxis versus concizumab prophylaxis.
  Interventions: Drug: Concizumab
- Arm 3: Concizumab prophylaxis (Experimental): The HA patients enrolled into the concizumab phase 2 trial NN7415-4255 (explorer 5) will be offered enrolment into this arm.
  Interventions: Drug: Concizumab
- Arm 4: Concizumab prophylaxis (Experimental): Arm 4 will include patients previously on prophylaxis with factor products with a minimum of 24 weeks observation in NN7415-4322 (explorer 6) (at least 30 HA and 30 HB patients).
  In addition, arm 4 will also include: 1) Patients who were randomised to arms 1 and 2 before the treatment pause. 2) HA patients who were in NN7415-4255 (explorer 5) at the time of the treatment pause, and who have now completed explorer 5. 3) On demand patients included after arms 1 and 2 are closed.
  Interventions: Drug: Concizumab

INTERVENTIONS:
Drug: Concizumab — When patients are randomised/allocated to concizumab prophylaxis, they will receive a loading dose of 1.0 mg/kg concizumab at visit 2a (week (Wk) 0) (arm 2, 3 and 4) or visit 9a (Wk 24) (arm 1) followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week dose adjustment period on 0.20 mg/kg concizumab, the patients can be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab. A potential dose adjustment will take place at visit 4a.1 (Wk 6) or 9a.3 (Wk 30) and will be based on the concizumab exposure level measured at the previous visit 4a (Wk 6) or 9a.2 (Wk 28). Patients who have concizumab exposure levels of 200-4000 ng/mL will stay at 0.20 mg/kg concizumab. Patients in arm 1 will continue on-demand treatment with their usual replacement therapy until visit 9a (week 24; end of main part). In the extension part, patients in arm 1 will receive daily concizumab subcutaneous injections.

SUMMARY:
This study will test how well a new medicine called concizumab works in the body of people with haemophilia A or B without inhibitors. The purpose is to show that concizumab can prevent bleeds in the body and is safe to use. Participants who usually only take medicine to treat bleeds (on-demand) will be placed in one of two groups. In one group participants will get study medicine from the start of the study. In the other group participants will continue with their normal medicine and get study medicine after 6 months. Which treatment the participant gets is decided by chance. Participants who usually take medicine to prevent bleeds (prophylaxis treatment) or who are already being treated with concizumab (study medicine) will receive the study medicine from the start of the study. Participants will have to inject themselves with the study medicine 1 time every day under the skin. This can be done at home. The study doctor will hand out the medicine in the form of a pen-injector. The pen-injector will contain the study medicine. The study will last for up to 8 years. The length of time the participant will be in the study depends on when they agreed to take part and when the medicine is available for purchase in their country (or 31 December 2027 at the latest). The time between visits will be approximately 4 weeks for the first 6 to 12 months depending on the group participants are in, and approximately 8 weeks for the rest of the study. If the participant attends extra visits due to the prescription medicine not being available for purchase in their country, these will be 14 weeks apart. Participants will be asked to record information in an electronic diary during the study and may also be asked to wear an activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male aged 12 years or older at the time of signing informed consent.
* Congenital severe haemophilia A (FVIII below 1%) or B (FIX equal to or below 2%).

Exclusion Criteria:

* Known or suspected hypersensitivity to any constituent of the trial product or related products.
* Known inherited or acquired coagulation disorder other than congenital haemophilia.
* Presence of confirmed inhibitors 0.6 BU or greater at screening.
* History of thromboembolic disease (includes arterial and venous thrombosis including myocardial infarction, pulmonary embolism, cerebral infarction/thrombosis, deep vein thrombosis, other clinically significant thromboembolic events and peripheral artery occlusion). Current clinical signs of, or treatment for thromboembolic disease. Patients who in the judgement of the investigator are considered at high risk of thromboembolic events (thromboembolic risk factors could include, but are not limited to, hypercholesterolemia, diabetes mellitus, hypertension, obesity, smoking, family history of thromboembolic events, arteriosclerosis, other conditions associated with increased risk of thromboembolic events.)

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2028-02-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (107):
- United States (12):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Center for Inherited Blood Disorders, Orange, California
  - Center for Blood Disorders Augusta University, Augusta, Georgia
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - University of Iowa_Iowa City, Iowa City, Iowa
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, Lansing, Michigan
  - Novant Hlth Vasc Ins Charlotte, Charlotte, North Carolina
  - M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center_Nashville_0, Nashville, Tennessee
  - University of Texas San Antonio, San Antonio, Texas
  - Versiti, CCBD, Milwaukee, Wisconsin
- Algeria (2):
  - Haematology and Blood Bank Department, Algiers
  - CHU Constantine BEN BADIS/ Hematology department, Constantine
- Australia (3):
  - The Alfred, Melbourne, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Fiona Stanley Hospital - Haemophilia and Haemostasis Centre, Murdoch, Western Australia
- University Clinical Center of Republic Srpska (205), Banja Luka, Bosnia and Herzegovina
- Bulgaria (2):
  - UMHAT Tsaritsa Yoanna-ISUL EAD, Sofia
  - UMHAT "Sveta Marina" EAD Clinic of Pediatric Clinical Hemat, Varna
- Canada (2):
  - Eastern Health Authority, St. John's, Newfoundland and Labrador
  - Hamltn Hth Sci/McMstr Child Hosp, Hamilton, Ontario
- KBC Zagreb, Rebro, Hemofilija centar, Zagreb, Croatia
- Copenhagen Center for Heamatology, Copenhagen, Denmark
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (6):
  - Centre Hospitalier Regional Et Universitaire de Brest-Hopital de La Cavale Blanche, Brest
  - CHU de Caen - Côte de Nacre, Caen
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Nantes-Hopital Hotel-Dieu, Nantes
  - Hôpital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Saint Etienne-Hopital Nord, Saint-Priest-en-Jarez
- Germany (2):
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
  - Universitätsklinikum des Saarlandes - Hämostaseologie und Transfusionsmedizin, Homburg
- MH Eü. Központ -Orszagos Haemophilia Kozpont, Budapest, Hungary
- India (5):
  - St. John's Medical college and Hospital, Bangalore, Karnataka
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - J K Lon Hospital, Jaipur, Rajasthan
  - CMCV, Ranipet, Tamil Nadu
- Sheba MC The Israeli National Hemophilia Center, Tel Litwinsky, Israel
- Italy (4):
  - Dipartimento di Ematologia Univ. Firenze, Florence, FI
  - Istituto di Medicina Int. A. Bianchi Bonomi Univ. Milano, Milan, MI
  - Policlinico Umberto I Sezione Ematologia, Roma
  - A.O.U Città Salute Scienza Torino, Torino
- Japan (11):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Hiroshima University Hospital, Hematology, Hiroshima
  - Hyogo prefectural kobe children's hospital, Hyōgo
  - Itoigawa sogo Hospital_Department of Pediatrics, Niigata
  - Osaka National Hospital, Osaka
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Saitama Medical Univ. Hospital, Saitama
  - Shizuoka Children's Hospital, Hematology-Oncology, Shizuoka
  - Shizuoka Children's Hospital, Shizuoka
  - National Center for Child Health and Development_Hematology, Tokyo
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- Lithuania (2):
  - Children Oncohaematology department Children's Hospital,, Vilnius
  - Vilnius University hospital Santaros klinikos, Vilnius
- Hospital Ampang, Ampang, Selangor, Malaysia
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico
- Poland (6):
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki, Oddzial Kliniczny Hematologii, Krakow, Lesser Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 1 Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
  - Uniwersytecki Szpital Dzieciecy, Dzial Krwiolecznictwa, Lublin
  - Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego We Wroclawiu, Wroclaw
- ULS São João, E.P.E., Porto, Portugal
- Russia (5):
  - Children Regional Clinical Hospital, Krasnodar
  - Morozovskaya municipal children hospital, Moscow
  - National Medical Research institution of haemotology, Moscow
  - Republican Hospital n.a. V. A. Baranov, Petrozavodsk
  - City out-patient clinic 37, City Hemophilia Centre, Saint Petersburg
- Serbia (4):
  - Clinical Centre of Serbia, Institute for Haematology, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
  - University Clinical Centre Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
- Nemocnica sv. Cyrila a Metoda, UNB,Klinika hemat. a transfuz, Bratislava, Slovakia
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
  - Pietersburg Hospital, Polokwane, Limpopo
- South Korea (5):
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Daejeon Eulji University Hospital, Daejeon
  - Jeju National University Hospital, Jeju City
  - Jeju National University Hospital, Jeju-do
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Univ. Central de Asturias, Oviedo
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
- Sweden (2):
  - Koagulationsmottagning, Malmo
  - Koagulationsmottagningen, Solna
- Universitätsspital Zürich - Klinik für Medizinische Onkologie und Hämatologie, Zurich, Switzerland
- RAMA -Hemato-Med_Department of Haematology, Bangkok, Thailand
- Turkey (Türkiye) (9):
  - Gazi University, Ankara, Beşevler/Ankara
  - Gazi Üniversitesi Hastanesi- Hematoloji, Ankara, Beşevler/Ankara
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Onkoloji Enstitüsü, Capa-ISTANBUL, Capa-ISTANBUL
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Hacettepe Üniversitesi Hastanesi- Endokrinoloji, Ankara
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi-Hematoloji, Edirne
  - Ege Üniversitesi Hastanesi- Hematoloji, Izmir
  - Ondokuz Mayis University Medical Faculty Ped. Haematology, Samsun
- Ukraine (2):
  - National specialized children's hospital 'OHMATDYT' - Haemostasis centre, Kyiv
  - Institute of blood pathology and transfusion medicine of NAMSU - General and haematol. surgery, Lviv
- United Kingdom (4):
  - Belfast City Hospital, Belfast
  - Royal Free Haemophilia Comprehensive Care Center, London
  - Royal Free Haemophilia Comprehensive Care Centre, London
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Angchaisuksiri P, von Mackensen S, Apte S, Benson G, Eichler H, Findley A, Matsushita T, Mazini Tavares CM, Puggaard Ravn M, Sathar J, Villarreal Martinez L, Young G. Concizumab prophylaxis in people with hemophilia A or B without inhibitors: patient-reported outcome results from the phase 3 explorer8 study. Res Pract Thromb Haemost. 2025 Feb 20;9(2):102705. doi: 10.1016/j.rpth.2025.102705. eCollection 2025 Feb. PMID 40166710
- [Derived] Chowdary P, Angchaisuksiri P, Apte S, Astermark J, Benson G, Chan AKC, Jimenez Yuste V, Matsushita T, Hogh Nielsen AR, Sathar J, Sutton C, Saulyte Trakymiene S, Tran H, Villarreal Martinez L, Wheeler AP, Windyga J, Young G, Thaung Zaw JJ, Eichler H. Concizumab prophylaxis in people with haemophilia A or haemophilia B without inhibitors (explorer8): a prospective, multicentre, open-label, randomised, phase 3a trial. Lancet Haematol. 2024 Dec;11(12):e891-e904. doi: 10.1016/S2352-3026(24)00307-7. Epub 2024 Nov 6. PMID 39521008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 68 sites in 31 countries.
Pre-assignment Details: Data is reported till cutoff date 27-Dec-2022 and study is still ongoing. Initially, participants were randomised to arm 1 or 2 or to non-randomised arms 3 or 4. There was a treatment pause due to investigation of thromboembolic events. After treatment pause, participants randomised to arms 1 or 2 before pause entered arm 4. Participants allocated to arms 3 and 4 before pause re-entered arms initially allocated to. New participants were randomized in arms 1and 2.
Groups:
- Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA: Participants with HA received their on-demand treatment for a minimum of 24 weeks. After treatment pause, participants initially randomised to arm 1 were to enter arm 4. Subsequently, following the main phase, participants transitioned to the new dosing regimen for concizumab and were scheduled to undergo concizumab prophylaxis in the trial's extension phase.
- Extension Phase Arm 1: Concizumab PPX - Participants With HA: Participants with HA who completed the main part were offered concizumab PPX in the extension part for up to an additional 353 weeks.
- Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA: Participants with HA received a loading dose of 1.0 milligrams per kilograms (mg/kg) concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg. After treatment pause, participants initially randomised to arm 2 were to enter arm 4.
- Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA: Participants with HA received a loading dose (participants entering from the phase 2 trial [N7415-4255] (NCT03196297) were not to receive a loading dose) of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg.
- Arm 4: Concizumab PPX - Participants With HA: Participants with HA previously on PPX with factor products and a minimum of 24 weeks of observation in the non interventional study 4322 (NCT03741881) were allocated to Arm 4. Additionally, Arm 4 also included participants who were randomised to arms 1 (no PPX) and 2 (concizumab PPX) before the treatment pause, participants who were in the phase 2 trial 4255 at the time of the treatment pause, and who had subsequently completed the trial when concizumab treatment was restarted and on-demand participants included after arms 1 and 2 were closed. The original dosing regimen was a loading s.c. dose of 1.0 mg/kg concizumab on the first day of treatment, followed by a maintenance dose of 0.25 mg/kg concizumab given as a daily s.c. injection from the second day and onwards. After the concizumab treatment pause and the treatment restart, participants received a loading dose of 1.0 mg/kg concizumab at visit 2a followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could have their dose increased to 0.25 mg/kg or decreased to 0.15 mg/kg concizumab or they could remain at a dose of 0.20 mg/kg.
- Arm 1: Previous OnD Treatment: No PPX - Participants With HB: Participants with HB received their on-demand treatment for a minimum of 24 weeks. After treatment pause, participants initially randomised to arm 1 were to enter arm 4. Subsequently, following the main phase, participants transitioned to the new dosing regimen for concizumab and were scheduled to undergo concizumab prophylaxis in the trial's extension phase.
- Extension Phase Arm 1: Concizumab PPX - Participants With HB: Participants with HB who completed the main part were offered concizumab PPX in the extension part for up to an additional 353 weeks.
- Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB: Participants with HB received a loading dose of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg. After treatment pause, participants initially randomised to arm 2 were to enter arm 4.
- Arm 4: Concizumab PPX - Participants With HB: Participants with HB previously on PPX with factor products and a minimum of 24 weeks of observation in the non interventional study 4322 (NCT03741881) were allocated to Arm 4. Additionally, Arm 4 also included participants who were randomised to arms 1 (no PPX) and 2 (concizumab PPX) before the treatment pause, participants who were in the phase 2 trial 4255 at the time of the treatment pause, and who had subsequently completed the trial when concizumab treatment was restarted and on-demand participants included after arms 1 and 2 were closed. The original dosing regimen was a loading s.c. dose of 1.0 mg/kg concizumab on the first day of treatment, followed by a maintenance dose of 0.25 mg/kg concizumab given as a daily s.c. injection from the second day and onwards. After the concizumab treatment pause and the treatment restart, participants received a loading dose of 1.0 mg/kg concizumab at visit 2a followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could have their dose increased to 0.25 mg/kg or decreased to 0.15 mg/kg concizumab or they could remain at a dose of 0.20 mg/kg.
Period: Main Part (Before the Treatment Pause)
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB
Started | 1 | 0 | 3 | 10 | 18 | 1 | 0 | 2 | 2
Completed | 0 (Participant discontinued from arm 1 was allocated to arm 4, however was not exposed to concizumab treatment in arm 4- concizumab PPX: participants with HA. This participant was included in the safety analysis set (SAS).) | 0 | 2 | 9 | 13 | 1 | 0 | 2 | 2
Not Completed | 1 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Main Part (After the Treatment Pause)
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB
Started | 9 | 0 | 18 | 9 | 46 (Participants restarting from before treatment pause = 13 Participants moved from old arm 1+2 = 2 (0+2) Participants allocated after restart = 31) | 12 | 0 | 24 | 30 (Participants restarting from before treatment pause = 2 Participants moved from old arm 1+2 = 3 (1+2) Participants allocated after restart = 25)
Completed | 7 | 0 | 17 | 6 | 45 | 10 | 0 | 23 | 25
Not Completed | 2 | 0 | 1 | 3 | 1 | 2 | 0 | 1 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 5
Not completed — Unspecified reason | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Extension Part
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB
Started | 0 | 7 | 17 | 6 | 45 | 0 | 10 | 23 | 25
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 7 | 17 | 6 | 45 | 0 | 10 | 23 | 25
Not completed — Ongoing | 0 | 7 | 17 | 6 | 45 | 0 | 10 | 23 | 25

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analysed based on the on-treatment without data before restart (OTexBR) analysis set. OTexBR analysis data set was defined as the observation period after the restart of treatment where participants were considered to be affected by no PPX (on-demand treatment) or concizumab PPX with the new concizumab dosing regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HB | Total
Number analyzed (Participants) | 9 | 12 | 18 | 24 | 9 | 46 | 30 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.7 (21.3) | 30.4 (17.5) | 30.7 (9.6) | 28.0 (12.0) | 43.7 (18.0) | 30.4 (13.4) | 31.6 (13.3) | 31.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 9 | 12 | 18 | 24 | 9 | 46 | 30 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 2 | 4 | 3 | 12
  Not Hispanic or Latino | 8 | 11 | 18 | 23 | 7 | 41 | 27 | 135
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Asian | 1 | 6 | 8 | 10 | 3 | 13 | 1 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4
  White | 7 | 6 | 9 | 12 | 6 | 30 | 27 | 97
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Haemophilia A Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Bleeding Episodes
Description: Rate of treated spontaneous and traumatic bleeding episodes for haemophilia A participants without inhibitors is presented. The observation period used for reporting this endpoint is on-treatment without ancillary therapy excluding data before restart (OTwoATexBR). It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of annualised bleeding rate (ABR). Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen. Confirmatory analyses cut-off was defined as when all participants on no PPX (arm 1) had completed the 24-week visit or withdrawn and all participants on concizumab PPX (in arms 2 and 4) had completed the 32-week visit or withdrawn.
Time Frame: On demand (arm 1): From week 0 up until start of concizumab treatment (week 24); Concizumab (arm 2): From week 0 up until the confirmatory analyses cut-off
Population: FAS included all participants randomised to the new concizumab PPX dosing regimen or on-demand treatment after the treatment pause or allocated to arm 3 or 4 with the new concizumab PPX dosing regimen. This endpoint is only defined for arms 1 and 2 as per protocol.
Measure: Median (Inter-Quartile Range); unit: Events per year
Groups:
- Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA: Participants with HA received a loading dose of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg. After treatment pause, participants initially randomised to arm 2 were to enter arm 4.
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA
Number analyzed (Participants) | 9 | 18
Events per year | 19.6 [17.3 to 30.4] | 2.9 [0.0 to 5.2]
Statistical Analysis 1: Comparison: Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA vs Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA; Test type: Superiority — Bleeding endpoints were analysed using a negative binomial regression model with the logarithm of the length of the observation period included (in years) as offset with treatment and bleeding frequency prior to screening as factors; p < 0.001, Negative binomial regression; ABR ratio = 0.14, 95% CI 2-sided [0.07 to 0.29]

2. Primary Outcome: Haemophilia B Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Bleeding Episodes
Description: Rate of treated spontaneous and traumatic bleeding episodes for haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen. Confirmatory analyses cut-off was defined as when all participants on no PPX (arm 1) had completed the 24-week visit or withdrawn and all participants on concizumab PPX (in arms 2 and 4) had completed the 32-week visit or withdrawn.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 12 | 24
Events per year | 14.9 [3.3 to 22.1] | 1.6 [0.0 to 4.8]
Statistical Analysis 1: Comparison: Arm 1: Previous OnD Treatment: No PPX - Participants With HB vs Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Negative binomial regression; ABR ratio = 0.21, 95% CI 2-sided [0.10 to 0.45]

3. Secondary Outcome: Haemophilia A Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Bleeding Episodes
Description: Rate of treated spontaneous and traumatic bleeding episodes for haemophilia A participants without inhibitors in arm 4 participants who had been on stable PPX at least 24 weeks in study 4322 is presented. The observation period used for reporting this endpoint is on stable treatment without ancillary therapy excluding data before restart (OT stable woATexBR). It is defined as the time period where participants are on stable PPX in study NN7415-4322 combined with the time period after the treatment pause in NN7415-4307 where the same participants are on the maintenance dose and have not used factor-containing products not related to treatment of a bleed. The data is reported in the terms of ABR.
Time Frame: For previous PPX (study 4322): After an initial period on PPX treatment of at least 24 weeks until end of study (maximum 115 weeks) For concizumab PPX (trial 4307): After an initial 5-8 weeks dose adjustment period and up until 56 week cut off
Population: Intra-participant analysis set (IPAS) included participants in arm 4 that were on a stable PPX regimen for at least 24 weeks in NN7415-4322 and who entered the maintenance period in this trial NN7415-4307. The participants reported in both arms/groups represent the same 29 participants, with results reported from Study 4322 and this study (Study 4307). The endpoint is only defined for arm 4 (previous PPX-study 4322) and arm 4 (concizumab PPX-study 4307) as per protocol.
Measure: Median (Inter-Quartile Range); unit: Events per year
Groups:
- Arm 4: Previous PPX (Study 4322) - Participants With HA: Arm 4 participants with haemophilia A who were on stable PPX for atleast 24 weeks in study 4322 and continued till end of study (until 115 weeks).
- Arm 4: Concizumab PPX (Study 4307) - Participants With HA: Arm 4 participants with haemophilia A who were on stable PPX for atleast 24 weeks in study 4322 and who entered the maintenance period in 4307.
Arm/Group | Arm 4: Previous PPX (Study 4322) - Participants With HA | Arm 4: Concizumab PPX (Study 4307) - Participants With HA
Number analyzed (Participants) | 29 | 29
Events per year | 2.2 [0.8 to 6.2] | 1.7 [0.5 to 4.8]

4. Secondary Outcome: Haemophilia B Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Bleeding Episodes
Description: Rate of treated spontaneous and traumatic bleeding episodes for haemophilia B participants without inhibitors in arm 4 participants who had been on stable PPX at least 24 weeks in study 4322 is presented. The observation period used for reporting this endpoint is OT stable woATexBR. It is defined as the time period where participants are on stable PPX in study NN7415-4322 combined with the time period after the treatment pause in NN7415-4307 where the same participants are on the maintenance dose and have not used factor-containing products not related to treatment of a bleed. The data is reported in the terms of ABR.
Time Frame: as for outcome 3
Population: IPAS included participants in arm 4 that were on a stable PPX regimen for at least 24 weeks in NN7415-4322 and who entered the maintenance period in this trial NN7415-4307. The participants reported in both arms/groups represent the same 29 participants, with results reported from Study 4322 and this study (Study 4307). The endpoint is only defined for arm 4 (previous PPX-study 4322) and arm 4 (concizumab PPX-study 4307) as per protocol.
Measure: Median (Inter-Quartile Range); unit: Events per year
Groups:
- Arm 4: Previous PPX (Study 4322) - Participants With HB: Arm 4 participants with haemophilia B who were on stable PPX for atleast 24 weeks in study 4322 and continued till end of study (until 115 weeks).
- Arm 4: Concizumab PPX (Study 4307) - Participants With HA: Arm 4 participants with haemophilia B who were on stable PPX for atleast 24 weeks in study 4322 and who entered the maintenance period in 4307.
Arm/Group | Arm 4: Previous PPX (Study 4322) - Participants With HB | Arm 4: Concizumab PPX (Study 4307) - Participants With HA
Number analyzed (Participants) | 22 | 22
Events per year | 2.1 [0.9 to 4.2] | 1.3 [0.0 to 6.4]

5. Secondary Outcome: Haemophilia A Participants Without Inhibitors: Rate of Treated Spontaneous Bleeding Episodes
Description: Rate of treated spontaneous bleeding episodes for haemophilia A participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: On demand (arm 1): From randomisation after the pause (week 0) up until start of concizumab treatment (week 24) Concizumab (arm 2): From start of the new concizumab dosing regimen (week 0) up until the 56 week cut-off
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Groups:
- Arm 2: Concizumab PPX - Participants With HA: Participants with HA received a loading dose of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg. After treatment pause, participants initially randomised to arm 2 were to enter arm 4.
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Concizumab PPX - Participants With HA
Number analyzed (Participants) | 9 | 18
Events per year | 19.3 [7.2 to 20.5] | 1.0 [0.0 to 3.6]

6. Secondary Outcome: Haemophilia B Participants Without Inhibitors: Rate of Treated Spontaneous Bleeding Episodes
Description: Rate of treated spontaneous bleeding episodes for haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 12 | 24
Events per year | 10.8 [3.3 to 17.8] | 1.0 [0.0 to 2.5]

7. Secondary Outcome: Haemophilia A Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Joint Bleeding Episodes
Description: Rate of treated spontaneous and traumatic joint bleeding episodes for haemophilia A participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Concizumab PPX - Participants With HA
Number analyzed (Participants) | 9 | 18
Events per year | 13.0 [10.7 to 28.3] | 2.0 [0.0 to 4.0]

8. Secondary Outcome: Haemophilia B Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Joint Bleeding Episodes
Description: Rate of treated spontaneous and traumatic joint bleeding episodes for haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 12 | 24
Events per year | 10.0 [3.3 to 18.0] | 2.0 [0.0 to 3.7]

9. Secondary Outcome: Haemophilia A Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Target Joint Bleeding Episodes
Description: Rate of treated spontaneous and traumatic target joint bleeding episodes for haemophilia A participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Concizumab PPX - Participants With HA
Number analyzed (Participants) | 9 | 18
Events per year | 4.3 [1.6 to 13.0] | 1.7 [0.0 to 3.0]

10. Secondary Outcome: Haemophilia B Participants Without Inhibitors: Rate of Treated Spontaneous and Traumatic Target Joint Bleeding Episodes
Description: Rate of treated spontaneous and traumatic target joint bleeding episodes for haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTwoATexBR. It is defined as the time period after the restart where participants are treated by concizumab treatment or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleeding episode. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 12 | 24
Events per year | 2.2 [0.0 to 8.1] | 0.7 [0.0 to 1.5]

11. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Thromboembolic Events
Description: Number of thromboembolic events in haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is on-treatment (OT). It is defined as the time period where participants were considered to be affected by no PPX (on-demand treatment) or concizumab PPX. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: On demand (arm 1): from week 0 until start of concizumab treatment (week 24). Concizumab (arms 2-4): From week 0 up until the 56 week cut-off. Concizumab (arm 1 extension part): From start of concizumab treatment (week 25) up until the 56 week cut-off
Population: SAS was defined as all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analysed = Participants with available data for the outcome measure. The endpoint is applicable for reported arms [for participants with HA (arm1, arm 2, arm 3, arm 4, arm 1 extension part) and participants with HB (arm 1, arm 2, arm 4, arm 1 extension part)] only.
Measure: Number; unit: Events
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 9 | 18 | 10 | 52 | 7 | 12 | 24 | 30 | 10
Events | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Thromboembolic Events
Time Frame: From week 0 to end of trial (up to 384 weeks)
Reporting Status: Not Posted, anticipated posting 2028-12

13. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Hypersensitivity Type Reactions
Description: Number of hypersensitivity type reactions in haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OT. It is defined as the time period where participants were considered to be affected by no PPX (on-demand treatment) or concizumab PPX. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: Reactions
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 9 | 18 | 10 | 52 | 7 | 12 | 24 | 30 | 10
Reactions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Hypersensitivity Type Reactions
Time Frame: From week 0 to end of trial (up until 384 weeks)
Reporting Status: Not Posted, anticipated posting 2028-12

15. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Injection Site Reactions
Description: Number of injection site reactions in haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OT. It is defined as the time period where participants were considered to be affected by no PPX (on-demand treatment) or concizumab PPX. Week 0 is defined as time of randomisation to on-demand administration after the pause or time of start of the new concizumab dosing regimen.
Time Frame: On demand (arm 1 main part): from randomisation (week 0) until start of concizumab treatment (week 24). Concizumab (arms 2-4): From week 0 up until the 56 week cut-off. Concizumab (arm 1 extension part): From week 25 up until the 56 week cut-off
Population: as for outcome 11
Measure: Number; unit: Reactions
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB
Number analyzed (Participants) | 9 | 18 | 10 | 52 | 7 | 12 | 24 | 30 | 10
Reactions | 0 | 1 | 0 | 14 | 1 | 0 | 2 | 28 | 0

16. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Injection Site Reactions
Time Frame: From week 0 to end of trial (up until 384 weeks)
Reporting Status: Not Posted, anticipated posting 2028-12

17. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Participants With Antibodies to Concizumab
Time Frame: Concizumab (arms 2-4): From start of concizumab treatment (week 0) up until the 56 week cut-off. Concizumab (arm 1 extension part): From start of concizumab treatment (week 25) up until the 56 week cut-off
Reporting Status: Not Posted, anticipated posting 2028-05

18. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Number of Participants With Antibodies to Concizumab
Time Frame: From week 0 to end of trial (up until 384 weeks)
Reporting Status: Not Posted, anticipated posting 2028-12

19. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Pre-dose (Trough) Concizumab Plasma Concentration (Ctrough)
Description: Ctrough for haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is on-treatment without data before re-start (OTexBR). It is defined as the time period after restart where participants were considered to be affected by no PPX (on-demand treatment) or treatment with the new concizumab regimen.
Time Frame: Pre-dose (prior to the concizumab administration at week 24)
Population: SAS was defined as all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analysed = Participants with available data for the outcome measure. The endpoint is applicable for reported arms [for participants with HA (arm 2, arm 3, arm 4) and participants with HB (arm 2, arm 4)] only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HA: Participants with HA who were on a stable PPX regimen for at least 24 weeks in study 4322 and who entered the maintenance period in the present trial, who were randomised to arms 1 (no PPX) and 2 (concizumab PPX) before the treatment pause, participants who were in the phase 2 trial 4255 at the time of the treatment pause, and who had subsequently completed the trial when concizumab treatment was restarted and on-demand participants included after arms 1 and 2 were closed were all allocated to Arm 4 and received a loading dose of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg.
- Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB: Participants with HB received a loading dose of 1.0 milligrams per kilograms (mg/kg) concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg. After treatment pause, participants initially randomised to arm 2 were to enter arm 4.
- Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HB: Participants with HB who were on a stable PPX regimen for at least 24 weeks in study 4322 and who entered the maintenance period in the present trial, who were randomised to arms 1 (no PPX) and 2 (concizumab PPX) before the treatment pause, participants who were in the phase 2 trial 4255 at the time of the treatment pause, and who had subsequently completed the trial when concizumab treatment was restarted and on-demand participants included after arms 1 and 2 were closed were all allocated to Arm 4 and received a loading dose of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg.
Arm/Group | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HB
Number analyzed (Participants) | 15 | 7 | 45 | 23 | 26
nanograms per milliliter (ng/mL) | 767.7 (112.4) | 612.3 (274.9) | 729.3 (158.6) | 413.6 (234.7) | 719.7 (189.7)

20. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Pre-dose Thrombin Peak
Description: Pre-dose thrombin peak for haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTexBR. It is defined as the time period after restart where participants were considered to be affected by no PPX (on-demand treatment) or treatment with the new concizumab regimen.
Time Frame: Pre-dose (prior to the concizumab administration at week 24)
Population: SAS was defined as all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analysed = Participants with available data for the outcome measure. The endpoint is applicable for reported arms [for participants with HA (arm 1, arm 2, arm 3, arm 4) and participants with HB (arm 1, arm 2, arm 4)] only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HB
Number analyzed (Participants) | 7 | 15 | 7 | 43 | 9 | 22 | 26
nanomoles per liter (nmol/L) | 19.9 (117.7) | 98.3 (53.3) | 92.3 (69.0) | 92.1 (57.8) | 9.6 (110.7) | 54.6 (111.9) | 79.4 (57.1)

21. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Pre-dose Free Tissue Factor Pathway Inhibitor (TFPI) Concentration
Description: Pre-dose free TFPI for haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTexBR. It is defined as the time period after restart where participants were considered to be affected by no PPX (on-demand treatment) or treatment with the new concizumab regimen.
Time Frame: Pre-dose (prior to the concizumab administration at week 24)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HB
Number analyzed (Participants) | 7 | 16 | 7 | 44 | 11 | 23 | 26
ng/mL | 70.1 (12.3) | 11.1 (74.8) | 15.9 (75.8) | 9.6 (87.9) | 88.1 (14.6) | 16.3 (130.3) | 10.5 (107.4)

22. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Maximum Concizumab Plasma Concentration (Cmax)
Description: Cmax for haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTexBR. It is defined as the time period after restart where participants were considered to be affected by no PPX (on-demand treatment) or treatment with the new concizumab regimen.
Time Frame: Pre-dose, Week 24: 3 hours (h), 6h, 9h, 24h
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HB
Number analyzed (Participants) | 10 | 5 | 36 | 11 | 22
ng/mL | 1158.2 (61.9) | 583.4 (282.2) | 1029.7 (130.9) | 689.2 (190.5) | 828.0 (111.2)

23. Secondary Outcome: Haemophila A and Haemophilia B Participants Without Inhibitors: Area Under the Concizumab Plasma Concentration-time Curve (AUC)
Description: AUC for haemophilia A and haemophilia B participants without inhibitors is presented. The observation period used for reporting this endpoint is OTexBR. It is defined as the time period after restart where participants were considered to be affected by no PPX (on-demand treatment) or treatment with the new concizumab regimen.
Time Frame: Pre-dose, Week 24: 3 hours (h), 6h, 9h, 24h
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX (IPAS) + Concizumab PPX (Others) - Participants With HB
Number analyzed (Participants) | 10 | 5 | 36 | 11 | 22
nanograms*hour/milliliter (ng*hr/mL) | 23582.5 (68.2) | 11082.7 (268.0) | 20355.6 (135.2) | 13020.5 (182.7) | 16191.8 (118.2)

ADVERSE EVENTS:
Time Frame: Up to week 56 cut-off
Description: Safety analysis set (SAS) included all participants exposed to concizumab prophylaxis (PPX) or randomised to on-demand treatment. All presented AEs were treatment emergent AEs (TEAEs). TEAEs were defined as AEs which initiated or worsened during the time period where participants were considered to be affected by on demand treatment or concizumab treatment.
Arm/Group | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA | Extension Phase Arm 1: Concizumab PPX - Participants With HA | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA | Arm 4: Concizumab PPX - Participants With HA | Arm 1: Previous OnD Treatment: No PPX - Participants With HB | Extension Phase Arm 1: Concizumab PPX - Participants With HB | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB | Arm 4: Concizumab PPX - Participants With HB
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/18 | 0/10 | 1/52 | 0/12 | 0/10 | 0/24 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 1/18 | 1/10 | 10/52 | 2/12 | 0/10 | 6/24 | 2/30
Other Adverse Events (participants affected / at risk) | 2/9 | 5/7 | 10/18 | 8/10 | 40/52 | 2/12 | 5/10 | 12/24 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA (N=9) | Extension Phase Arm 1: Concizumab PPX - Participants With HA (N=7) | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA (N=18) | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA (N=10) | Arm 4: Concizumab PPX - Participants With HA (N=52) | Arm 1: Previous OnD Treatment: No PPX - Participants With HB (N=12) | Extension Phase Arm 1: Concizumab PPX - Participants With HB (N=10) | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB (N=24) | Arm 4: Concizumab PPX - Participants With HB (N=30)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Previous On Demand (OnD) Treatment: No Prophylaxis (PPX) - Participants With HA (N=9) | Extension Phase Arm 1: Concizumab PPX - Participants With HA (N=7) | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HA (N=18) | Arm 3: Concizumab Non-naive: Concizumab PPX - Participants With HA (N=10) | Arm 4: Concizumab PPX - Participants With HA (N=52) | Arm 1: Previous OnD Treatment: No PPX - Participants With HB (N=12) | Extension Phase Arm 1: Concizumab PPX - Participants With HB (N=10) | Arm 2: Previous OnD Treatment: Concizumab PPX - Participants With HB (N=24) | Arm 4: Concizumab PPX - Participants With HB (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 14 (14) | 0 (0) | 0 (0) | 3 (3) | 9 (9)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device physical property issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 8 (8) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Fibrinolysis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (6)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (10)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (9) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin fragment 1.2 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There was a pause in the concizumab clinical development programme during the period from March to August 2020, while thromboembolic events were investigated. As of 19 March 2020, all participants on concizumab had stopped treatment and switched to another available treatment as per investigator's discretion. Based on the investigation, risk mitigation actions (including new concizumab dosing regimen) were implemented and trial protocols updated before resuming.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT04082429/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04082429/SAP_001.pdf